CLINICAL TRIAL: NCT02266563
Title: Imaging [18F]AV-1451 and [18F]AV-45 in Acute and Chronic Traumatic Brain Injury
Brief Title: Amyloid and Tauopathy PET Imaging in Acute and Chronic Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Samuel Gandy (Other)
Responsible Party: Sponsor-Investigator, Samuel Gandy, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: GCO 14-0732
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury; Chronic Traumatic Encephalopathy; Mild Cognitive Impairment
Keywords: Traumatic Brain Injury; Chronic Traumatic Encephalopathy; Mild Cognitive Impairment; PET imaging; tauopathy; amyloid
MeSH Terms: conditions — Brain Injuries, Traumatic; Chronic Traumatic Encephalopathy; Cognitive Dysfunction; Tauopathies; Alzheimer Disease | interventions — florbetapir; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Traumatic Brain Injury (TBI) Group: TBI subjects will have a history of one or more concussions and have a memory complaint and objective decline that is considered to be worse than others of the same age (in the absence of an acute medical event). Severity classifications of the subjects selected for past history of TBI will be based upon established criteria used in TBI research (i.e., traumatically induced physiologic disruption of brain function as indicated by at least one of the following: any period of loss of consciousness, any loss of memory for events immediately before or after the accident, any alteration in mental state at the time of the accident, focal neurologic deficits that may or may not be transient). TBI cases will be those with mTBI (single or multiple concussion). Most recent injury must have occurred at least 1 year prior to study enrollment.
  Interventions: Drug: Amyvid PET Scan; Drug: T807 PET scan
- Mild Cognitive Impairment (MCI) Group: MCI Subjects will have MMSE scores between 24-30 (inclusive), a CDR of 0.5, have no depression, no history of TBI, and no dementia.
  Interventions: Drug: Amyvid PET Scan; Drug: T807 PET scan
- Healthy Control Group: Healthy control subjects will have no self or informant-reported problems with cognition, no depression, no history of TBI, and no dementia.
  Interventions: Drug: Amyvid PET Scan; Drug: T807 PET scan

INTERVENTIONS:
Drug: Amyvid PET Scan — A thin line will be inserted into a vein in one arm for the injection of the tracer. Subjects will begin the Amyvid PET scan 50-60 minutes after the injection of the tracer, and scanned for about 20 minutes.
  Other Names: [F18] AV-45; Florbetapir; Amyvid
Drug: T807 PET scan — Scanning will begin 80 minutes after the injection of the tracer, and last for about 20 minutes.
  Other Names: [F18] AV-1451

SUMMARY:
The potential long-term effects of Traumatic Brain Injury (TBI) are poorly understood. Repeated concussions have been associated with an elevated incidence of Alzheimer's disease (AD) along with a reduced age of onset. As repetitive TBI has been studied, a syndrome has now been identified: chronic traumatic encephalopathy (CTE). There are growing concerns about the long-term neurologic consequences of head impact exposure from routine participation in contact sports (e.g., boxing, football). Brain autopsies of athletes with confirmed CTE have demonstrated tau-immunoreactive neurofibrillary tangles and neuropil threads (known as tauopathy). The relationship between exposure to repetitive head impact and the subsequent development of chronic neurodegenerative disease has not been established. Further, as the diagnosis of CTE (defined by the presence of tauopathy) is presently made after death at autopsy, clinical tools and biomarkers for detecting it remain to be defined.

With the advent of FDA-approved PET amyloid imaging, clinicians and researchers are now able to estimate plaque density in the brains of living patients. However, there are critical limitations to amyloid imaging. Current evidence suggests that markers of the presence and severity of tauopathy may be able to address these limitations. The study will utilize both [18F] Florbetapir and [18F]-T807 PET imaging to investigate amyloid and tau accumulation in subjects with a history of concussions. In order to determine whether problems with cognition and memory are seen within the populations defined for the study, the researchers will administer a core battery of neurocognitive testing. This battery will assess cognitive abilities commonly affected by TBI, including processing speed, reaction time, new problem-solving, executive functions, attention and concentration, and learning and memory. These tests, in conjunction with the imaging, will be able to determine whether regional brain activity is associated with specific cognitive problems. The researchers will obtain PET and neurocognitive data in 3 cohorts: subjects with a history of TBIs, subjects with mild cognitive impairment (MCI) and no TBI history, and healthy controls.

The investigators aim to determine whether individuals with TBI are on the same trajectory of neurodegenerative disease seen in AD or in CTE. Because of the overlap in clinical/cognitive and some behavioral symptoms in AD and CTE, an additional biomarker tool is needed to prevent misdiagnosis. Accurate diagnosis is crucial in order to provide patients with appropriate treatment.

DETAILED DESCRIPTION:
The study involves two days of study visits. Subjects will be given a copy of the consent form on the morning of their first visit, and sign consent in a private room at Mount Sinai before any research related procedures are conducted. Subjects will then be brought to the Hess Center for Science in Medicine for injection for the [18F] AV-45 (or Amyvid) PET scan. On the second visit, which is to be conducted the day after the first visit, subjects will have the [18F]AV-1451 (or T807) PET scan and complete the neuropsychological testing battery.

Both PET scans will be done entirely for the purpose of research. The scans will be read by nuclear medicine physicians and a clinical report will be sent to the PI. Any clinically relevant findings will be sent to the treating physician and will be communicated to patients. During both visits, subjects will be allowed time for meals and breaks between study procedures.

Details of procedures:

Amyvid PET scan: At the first visit, each participant will have an Amyvid PET scan. The scan involves use of a "tracer", which is a radioactive sugar-like substance. This type of PET scan involves a tracer called AV-45 (also known as Florbetapir, and by the trade name of Amyvid). It has been approved by the FDA for use in PET imaging. It binds to beta-Amyloid plaques that may or may not be present in the brain. Amyloid plaque is a sticky substance (protein) that accumulates in the brain in larger amounts in people who may have Alzheimer's disease. A thin line will be inserted into a vein in one arm for the injection of the tracer. Subjects will begin the Amyvid PET scan 50-60 minutes after the injection of the tracer, and scanned for about 20 minutes.

T807 PET scan: On the day of the second visit, each participant will have an [F18] AV-1451 PET scan, also known as a T807 PET scan. This type of PET scan is being studied by the FDA as a diagnostic tool. This PET scan involves a very similar procedure to the Amyvid PET scan the day before. Like the Amyvid scan, a thin line will be inserted into a vein in one arm for the injection of the AV-1451 radiotracer. This tracer binds to clusters of Tau protein inside the brain called neurofibrillary tangles. These tangles are associated with both Alzheimer's disease and memory problems that may be related to multiple head injuries or concussions. Scanning will begin 80 minutes after the injection of the tracer, and last for about 20 minutes.

Neuropsychological testing battery: The neuropsychological assessment is a battery of pencil and paper tests that measure memory and thinking abilities. In total it takes about two hours to complete.

ELIGIBILITY:
Inclusion Criteria:

* males between 40 to 85 years of age
* individuals who participated in contact sports (e.g., active and retired NFL players, NHL players, boxers, NCAA athletes) and other individuals (including but not limited to veterans, breachers, or law enforcement officials with multiple blast exposures) who all have a history of one or more concussions and have a memory or cognitive complaint
* individuals with Mild Cognitive Impairment (MCI) and no history of concussion or TBI
* healthy controls with no history of head injury and no current cognitive or memory problems
* all participants require a study partner, who is well acquainted with the participant, to answer questions either in person or over the telephone about the individuals' activities of daily living, and to corroborate cognitive problems and past history of brain injury

Exclusion Criteria:

* any significant neurological disease, such as Alzheimer's disease, Parkinson's disease, vascular dementia, Huntington's disease, Pick's disease, Lewy Body Dementia, frontotemporal dementia, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, or multiple sclerosis
* any significant systemic illness or unstable medical condition, including: uncontrolled diabetes mellitus, uncorrected hypothyroidism or hyperthyroidism, or systemic cancer
* a history of schizophrenia or psychosis, alcohol or substance abuse or dependence within the past 6 months
* clinically significant impairment of liver or renal function
* significant cerebrovascular disease
* impairment of visual or auditory acuity sufficient to interfere with completion of study procedures
* education level < 10 years
* any subjects with a history of risk factors for Torsades de Pointes, or subjects taking drugs known to prolong the QT interval
* subjects who have had 2 or more PET scans within the past year, or other significant exposure to radiation (i.e., radiation therapy)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited through the Mount Sinai's Alzheimer's Disease Research Center (ADRC), the Memory and Aging Center (MAC), Center for Cognitive Health (CCH), and the NFL Neurological Program at the Icahn School of Medicine at Mount Sinai.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Uptake of [18F]T807 in the brain | 2 years
  To quantitatively assess the uptake of [18F]T807, a marker of tangles of tau protein in the brain, using positron emission tomography (PET) in individuals with a history of head injury or mTBI, with Mild Cognitive Impairment, and in healthy controls. Differences in uptake between the three groups will be measured.

SECONDARY OUTCOMES:
Uptake of [18F]AV-45 in the brain | 2 years
  To quantitatively assess the uptake of [18F]AV-45 (also known as Amyvid), a marker of Amyloid plaques, using positron emission tomography (PET) in individuals with a history of head injury or mTBI, with Mild Cognitive Impairment, and in healthy controls. Differences in uptake between the three groups will be measured.
Neuropsychological data composite score | 2 years
  2. Determining the relationship between [18F]-T807 imaging and cognitive problems. Neuropsychological raw data will be standardized and converted to z-scores. Correlational analysis with imaging data will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Gandy, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Dara Dickstein, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States